CLINICAL TRIAL: NCT05725291
Title: First-in-Human, Phase 1 Study of AMT-116 in Patients With Advanced Solid Tumors
Brief Title: AMT-116 in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Multitude Therapeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMT-116-01
Record Dates: First submitted 2023-02-02; First posted 2023-02-13 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Advanced Solid Tumor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- AMT-116 Dose Escalation (Experimental)
  Interventions: Drug: AMT-116

INTERVENTIONS:
Drug: AMT-116 — Administered intravenously

SUMMARY:
This first-in-human study will evaluate the Maximum Tolerated Dose (MTD) / the Recommended Phase 2 Dose (RP2D), safety, tolerability, anti-tumor activity, pharmacokinetics, pharmacodynamics and immunogenicity of AMT-116, in Patients with Advanced Solid Tumors

ELIGIBILITY:
Key Inclusion Criteria:

* Patients must be willing and able to sign the ICF, and to adhere to the study visit schedule and other protocol requirements.
* Age ≥18 years (at the time consent is obtained).
* Patients with histologically confirmed, unresectable advanced solid tumor. Preferred tumor types include head and neck, non-small cell lung, esophageal, pancreatic, large cell lung, colorectal, cervical, breast, bladder, gastric, biliary tract, skin squamous cell, liver, and basal cell cancer.
* Patients who have undergone at least one systemic therapy and have radiologically or clinically determined progressive disease during or after most recent line of therapy, and for whom no further standard therapy is available, or who are intolerable to standard therapy.
* Patients must have at least one measurable lesion as per RECIST version 1.1.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
* Both male and female patients must agree to use effective contraceptive methods.
* Patients must have adequate organ function.
* Women of child-bearing potential (WCBP) must have a negative serum pregnancy test.
* Male patients must agree to use a latex condom, even if they had a successful vasectomy, while on study treatment and for at least 12 weeks after the last dose of the IMP.
* Male patients must agree not to donate sperm, and female patients must agree not to donate eggs, while on study treatment and for at least 12 weeks after the last dose of the IMP.
* Availability of tumour tissue sample (either an archival specimen or a fresh biopsy material) at screening.

Key Exclusion Criteria:

* Prior therapy with ADC based on Top1 inhibitor.
* Central nervous system (CNS) metastasis.
* Active or chronic skin disorder requiring systemic therapy.
* History of Steven's Johnson's syndrome or Toxic Epidermal Necrolysis syndrome.
* Active ocular conditions requiring treatment or close monitoring, including, but not limited to: macular degeneration, papilledema, active diabetic retinopathy with macular oedema, wet age-related macular degeneration requiring intravitreal injections, or uncontrolled glaucoma.
* Persistent toxicities from previous systemic anti-neoplastic treatments of Grade >1.
* Systemic anti-neoplastic therapy within five half-lives or 21 days, whichever is shorter, prior to first dose of the IMP.
* Radiotherapy to lung field at a total radiation dose of ≥20 Gy within 6 months, wide-field radiotherapy (e.g., > 30% of marrow-bearing bones) within 28 days.
* Major surgery (not including placement of vascular access device or tumor biopsies) within 28 days prior to the first dose of the IMP, or no recovery from side effects of such intervention.
* Prior allogeneic or autologous bone marrow transplantation.
* Significant cardiac disease, such as recent (within six months prior to first dose of the IMP) myocardial infarction or acute coronary syndromes (including unstable angina pectoris), congestive heart failure (New York Heart Association class III or IV), uncontrolled hypertension, uncontrolled cardiac arrhythmias.
* Pregnant or breast-feeding females.

Note: Other protocol defined Inclusion/Exclusion criteria apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2023-07-25 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase 2 Dose (RP2D) | Up to 24 months
  The RP2D will be determined using dose limiting toxicities (DLTs) and all other available study data
Maximum Tolerated Dose (MTD) | Up to 24 months
  The MTD will be determined using DLTs
Type, incidence and severity of Adverse Events | Up to 24 months
  Safety and tolerability profile assessed by the Common Terminology Criteria for Adverse Events v5.0

SECONDARY OUTCOMES:
Overall Response Rate (ORR) according to the Response Evaluation Criteria in Solid Tumors (RECIST) v1.1 | Up to 24 months
  Proportion of patients achieving Complete Response (CR) or Partial Response (PR)
Disease Control Rate (DCR) according to the RECIST v1.1 | Up to 24 months
  Proportion of patients achieving CR, PR or Stable Disease (SD)
Progression-free Survival (PFS) | Up to 24 months
  Time from date of start of treatment to date of the first progression or death, whichever occurs first.
Concentration of anti-drug antibodies (ADA) | Up to 24 months
  Immunogenicity profile characterized by concentration of ADAs
Maximum observed concentration (C[max]) | Up to 24 months
  Pharmacokinetic profile characterized by the maximum observed concentration (C[max]) of AMT-116
Area under the curve (AUC) | Up to 24 months
  Pharmacokinetic profile characterized by the area under the curve (AUC) of AMT-116
Terminal half-life (t[1/2]) | Up to 24 months
  Pharmacokinetic profile characterized by the terminal half-life (t[1/2]) of AMT-116
Time to maximum concentration (Tmax) | Up to 24 months
  Pharmacokinetic profile characterized by the time to maximum concentration (Tmax) of AMT-116

CONTACTS AND LOCATIONS:
Overall Officials: Jermaine Coward, Principal Investigator — ICON Cancer Centre
Locations (10):
- United States (2):
  - Sarah Cannon Research Institute, Denver, Colorado
  - Mary Crowley Cancer Research Centers, Dallas, Texas
- American Samoa (2):
  - University of California San Francisco Cancer Center, San Francisco, California
  - Carolina BioOncology Institute, LLC, Cary, North Carolina
- Australia (6):
  - Macquarie University Hospital, Sydney, New South Wales
  - ICON Cancer Centre, Brisbane, Queensland
  - Southern Oncology Clinical Research Unit, Adelaide, South Australia
  - Alfred Hospital, Victoria Park, Victoria
  - Austin Health, Victoria Park, Victoria
  - Cabrini Hospital, Victoria Park, Victoria

IPD SHARING:
Plan to Share IPD: No